CLINICAL TRIAL: NCT05977907
Title: Neoadjuvant Pembrolizumab and IO102-103 Prior to Curative-intent Surgical Care for Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Neoadjuvant Pembrolizumab and IO102-103 for Squamous Cell Carcinoma of the Head and Neck (SCCHN).
Acronym: KIEO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: IO Biotech (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J22106; IRB00362497 (Other: JHM IRB)
Record Dates: First submitted 2023-07-25; First posted 2023-08-07 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: All participants receive same dose of drug. One Cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Cohort (Experimental): Neoadjuvant Pembrolizumab ( 400mg IV infusion x1) + IO102-103 ( Subcutaneous injection weekly x6)
  Adjuvant Pembrolizumab ( 400 mg IV infusion Every 6 weeks x8) + IO102-103 ( Subcutaneous injection every 3 week x6 then every 6 weeks x5)
  Interventions: Drug: Pembrolizumab; Drug: IO102-103

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab is an investigational drug in this study
  Other Names: Keytruda
Drug: IO102-103 — IO102-103 is an investigational drug in this study.

SUMMARY:
This research is being done to see if it is safe to give investigational combination of study drugs (Pembrolizumab and IO102-103) before surgery to people with surgically resectable (removable) newly diagnosed or recurrent metastatic SCCHN. This will be done by watching participants closely for possible side effects from Pembrolizumab and IO102-103. In addition, participants will be monitored for any delays to their surgery due to the study drugs.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age on day of signing informed consent.
* Patients with non-bulky/non-bulky squamous cell carcinomas of the head and neck, with an indication for surgical therapy.

  1. Surgically resectable disease - generally that is T1N1-N2B, T2-4N0-N2b stage are generally eligible (AJCC 7th), however exceptions can be made after approval by the PI for surgically appropriate cases.
  2. If determined per tumor board that a low-volume/non-bulky tumor of another stage is appropriate for resection (e.g. small volume T4 with a small amount of bone invasion) such tumors may also be considered for this study if recommendation in tumor board is such.
* Be appropriate candidates for resection and curative intent therapy in general.
* Have a performance status of 0 or 1 on the ECOG Performance Scale.
* Consent to undergo biopsy from a newly obtained core or excisional biopsy of a tumor lesion before study drug administration, and during treatment. Biopsy in case of progressive disease is optional.
* Demonstrate adequate organ function
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

  1. Abstinence is considered an adequate contraception method.

Exclusion Criteria:

* A Women of child bearing potential (WOCBP) who has a positive urine pregnancy test within 72 hours prior to treatment allocation/registration . If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor
* Has received prior systemic anti-cancer therapy for HNSCC including investigational agents within 4 weeks of first dose of study treatment.
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non- Central nervous system (CNS) disease.
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug (including live COVID-19 vaccines). Administration of killed vaccines is allowed. Administration of messenger RNA (mRNA) or peptide vaccines (e.g., for COVID-19) is allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, low grade cancers that are not expected to impact life expectancy within the next 3 years and not impact interpretation of this study are allowed
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs), unless it is systemic steroid therapy equal or less than outlined in exclusion criteria 7.

Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement .

therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.

* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has a known history of Hepatitis B or Hepatitis C virus
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial as per assessment of the treating physician. Chronic managed disorders that are not clinically active are acceptable.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* Has had an allogenic tissue/solid organ transplant.
* Congestive heart failure , unstable angina, serious uncontrolled cardiac arrhythmia, a myocardial infarction within 6 months prior to study entry or a history of myocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-12-14 (Actual); Primary Completion 2026-10-16 (Estimated); Study Completion 2028-10-16 (Estimated)

PRIMARY OUTCOMES:
Pathologic Treatment Response rate | From neoadjuvant therapy to surgical resection, up to 6 weeks
  To determine rate of pathologic treatment response ≥50% (pTR-2) / immune-related pathologic response criteria (irPRC) ≥ 50% rate to neoadjuvant pembrolizumab plus IO102-IO103 in SCCHN

SECONDARY OUTCOMES:
Major Pathologic Response | From neoadjuvant therapy to surgical resection, up to 6 weeks
  To determine the rate of major pathologic response with the neoadjuvant treatment approach
Disease progression | From neoadjuvant therapy to surgical resection, up to 6 weeks
  To determine progression-free survival in patients treated with immunotherapy-based neoadjuvant therapy followed by surgical resection
Overall survival | From neoadjuvant therapy to surgical resection, up to 6 weeks
  To determine overall survival in patients treated with immunotherapy-based neoadjuvant therapy followed by surgical resection
Overall Safety | Up to 100 days after the last dose of study drug
  To determine the safety and feasibility of the proposed treatment approach including severe adverse events (SAEs), AEs related treatment/surgery delays, and treatment related mortality. AEs and other toxicities will be graded using NCI Common Terminology Criteria for Adverse Events 5.0 (CTCAE)
ctDNA in comparison to other neoadjuvant treatments | 5 years
  To determine circulating tumor DNA (ctDNA) ≥50% response rate compared to another anti-Programed Cell Death protein 1 (PD-1) treated neoadjuvant cohort

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, M.D., Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (5):
- United States (5):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Providence Cancer Institute, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No